CLINICAL TRIAL: NCT01974869
Title: The Effect of Anti-Tumor Necrosis Factor Agents on Surgical Stress Response in Inflammatory Bowel Disease Patients Undergoing Abdominal Surgery
Brief Title: Anti Tumor Necrosis Factor Alpha Agents and Surgical Stress Response
Status: Completed | Type: Observational
Sponsor: El-Hussuna, Alaa, M.D. (Individual)
Responsible Party: Principal Investigator, Alaa El-Hussuna, Consultant surgeon, El-Hussuna, Alaa, M.D.
Other Study IDs: a-TNF
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Surgery,Crohn's disease,Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Inflammatory bowel diseases-1: Treatment with anti-tumor necrosis factor alpha agents
  Interventions: Drug: Anti-tumor necrosis factor alpha agents
- Inflammatory bowel diseases-2: Controls

INTERVENTIONS:
Drug: Anti-tumor necrosis factor alpha agents — Treatment with biologics
  Other Names: Biologics
  Groups: Inflammatory bowel diseases-1

SUMMARY:
Background: The immunologic response to stress is regulated by the cytokines. Anti-Tumor Necrosis Factor-α agents are antibodies directed against a key cytokine in the process angiogenesis and collagen synthesis. It is not known whether they intervene with surgical stress response increasing the rate of postoperative complications.

Method: Un-blinded prospective, non-interventional cohort single centre study including all the patients with Crohn's disease and Ulcerative Colitis undergoing abdominal surgery. Immunological and endocrinological parameters will measured in blood samples taken from these patients before and after surgery. Power calculations showed that 17 patients in each arm are needed.

DETAILED DESCRIPTION:
The baseline patient characteristics will be evaluated based on pilot tested data extraction sheets. The assessment will include demographics, clinical data as well as laboratory work up. The Charlson morbidity index, will be used to assess co-morbidity, the Nutritional risk score (NRS) to assess nutrition status and the Harvey-Bradshaw index (HBI) to evaluate the activity of Crohn's disease. The duration of surgical procedure, along with the amount of blood transfused, will be recorded in all patients.

Laboratory variables

The following variables will be assessed based on previous evidence about their role in surgical stress response:

1. Immunological parameters: Tumor necrosis factor-alpha, interleukin-1, interleukin-6, interleukin-10, C reactive protein, and white blood cell counts.
2. Endocrinological parameters: plasma cortisol, growth hormone , adrenocorticotropic hormone, epinephrin and norepinephrine

ELIGIBILITY:
Inclusion Criteria:

Patients with Crohn disease, ulcerative colitis and indeterminate colitis undergoing elective abdominal surgery (laparoscopic or open)

Exclusion Criteria:

No patients will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Crohn disease, ulcerative colitis and indeterminate colitis undergoing elective abdominal surgery (laparoscopic or open)
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
changes in inflammatory cytokines | pre-operative, at time of induction of anaethesia, 6,24 and 48 hours after the operation
  Primary outcome measure is the change in inflammatory cytokines Tumor Necrosis Factor-alpha, interleukin -1, interleukin -6, interleukin -10

SECONDARY OUTCOMES:
30 postoperative day complications. | 30 days after operation
  Secondary outcome measure is 30 postoperative day complications.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El-Hussuna, Principal Investigator — Slagelse Hospital
Locations (4):
- Denmark (4):
  - Århus University Hospital, Aarhus
  - Slagelse Hospitals, Copenhagen
  - Køge Hospital, Køge
  - OUH, Odense

IPD SHARING:
Plan to Share IPD: Yes
To be planned

REFERENCES:
- [Derived] El-Hussuna A, Qvist N, Zangenberg MS, Langkilde A, Siersma V, Hjort S, Gogenur I. No effect of anti-TNF-alpha agents on the surgical stress response in patients with inflammatory bowel disease undergoing bowel resections: a prospective multi-center pilot study. BMC Surg. 2018 Nov 3;18(1):91. doi: 10.1186/s12893-018-0425-0. PMID 30390672